CLINICAL TRIAL: NCT05582018
Title: Pilot Study to Assess the Safety and Effectiveness of the Use of BioTraceIO 360 for PSM and Planning, Monitoring and Assessment of Liver Tissue Ablation Procedures
Brief Title: Safety and Effectiveness of BioTraceIO 360 for Planning, Monitoring and Assessment of Liver Tissue Ablation Procedures
Acronym: PANORAMA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Techsomed Medical Technologies LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CL000030
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma; Metastatic Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- BioTrace (Experimental): Use of the BioTraceIO 360 device for planning, monitoring and assessment of liver tissue ablations
  Interventions: Device: BioTraceIO 360

INTERVENTIONS:
Device: BioTraceIO 360 — Use of the device for planning, monitoring and assessment of liver tissue ablations

SUMMARY:
Pilot study planned to demonstrate the safety and effectiveness of the use of BioTraceIO 360 for Planning, Monitoring and Assessment of liver tissue ablation procedures

Multi-center (up to 5 investigational sites) prospective single-arm clinical investigation.

Sample size - 30 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled and indicated for standard-of-care liver tumor ablation for either hepatocellular carcinoma (HCC) or metastatic liver tumor(s) microwave (MW) energy.
* Patient must have at least one prior CT or CECT scan (up to 6 months before enrollment).
* Tumor must be visualized on at least one diagnostic imaging modality (MRI or contrast-enhanced CT).
* Single tumor, or multiple tumors only if the distance between the ablated tumor and all other tumors allows for distinct separation between the necrotic zones.
* Distance between the tumor and the edge of any previous necrotic zones allows for distinct separation between the necrotic zones.
* At least 21 years of age.
* Able and willing to give informed consent.

Additional inclusion criteria for subgroup:

* Single ablation, using a single ablation needle, per tumor.

Exclusion Criteria:

* Planned ablation includes adjunctive means other than MW energy (e.g., ethanol, hepatic artery embolization, etc.).
* Planned ablation includes the use of more than two ablation needles, per tumor
* Ablation area cannot be visualized and monitored continuously using ultrasound throughout the entire ablation procedure.
* Pregnant or breastfeeding.
* Patient judged unsuitable for study participation by the physician for any other reason.
* Currently participating in another clinical trial of an unapproved investigational device or drug that has not concluded the follow-up period.
* Unable or unwilling to give informed consent.

Additional exclusion criteria for subgroup:

* Liver tumor that cannot be ablated with a single ablation needle, according to the investigator's clinical opinion.
* Planned ablation includes repositioning and/or overlapping ablations using a single ablation needle.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Effectiveness | 1 year
  The percentage of patients for whom (1) probe(s) position suggestion provided by the BioTraceIO 360 device is in agreement with the planned probe(s) position, as determined by the physician without the use of the device, or (2) clinically feasible probe(s) positioning suggestion was provided by the BioTraceIO 360 device, in addition to the planned probe(s) position by the physician without the use of the device.
Safety | 1 year
  Incidence and severity of device-related adverse

SECONDARY OUTCOMES:
Planning Module | 1 year
  The proportion of subjects in whom the physician has made changes and/or reported increased confidence to the planned ablation procedure after using the BioTraceIO 360 Planning Module compared to without using it.
Monitoring Module | 1 year
  A non-validated qualitative assessment for the physician regarding confidence during the procedure without and with the use of BioTraceIO 360 Monitoring Module if they could have made clinical decisions based on the use of the device.
Assessment Module (1) | 1 year
  A non-validated qualitative assessment on whether there were subjects, in whom the physician indicated that they would have changed the procedure and/or follow-up decision if they could have made clinical decisions based on the visualization of the tumor compared to the necrosis, using the BioTraceIO 360 Assessment Module at the end of the procedure.

OTHER OUTCOMES:
Assessment Module (2) | 1 year
  A non-validated qualitative assessment on whether there were subjects, for whom the BioTraceIO 360 Assessment Module indicated an incomplete ablation of the target tissue, compared to follow up 1-month post-procedure imaging.
Accuracy | 1 year
  A paired comparison between the DICE similarity coefficient, assessed for BioTraceIO 360 as measured during the ablation procedure (T=0) and the tissue damage area based on 24-hours post-procedure imaging (T=24), to the DICE similarity coefficient, assessed between the tissue damage area based on immediately post-procedure imaging (T=0) and the tissue damage area based on 24-hours post-procedure imaging (T=24).
Sensitivity | 1 year
  Sensitivity of the BioTraceIO 360 at T=0 compared to imaging at T=24.
Precision | 1 year
  Precision of the BioTraceIO 360 at T=0 compared to imaging at T=24.

CONTACTS AND LOCATIONS:
Locations (1):
- Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No